CLINICAL TRIAL: NCT02175134
Title: IFN-gamma-releasing Assay Based Approach in Patients With Suspected Tuberculous Peritonitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment rate
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Han Kim, Associate Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2014-0616
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Suspected Tuberculous Peritonitis
Keywords: tuberculosis; peritonitis; laparoscopy
MeSH Terms: conditions — Tuberculosis; Peritonitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional diagnostic flow arm (No Intervention): Perform the laparoscopic biopsy as a discretion of attending physician's decision
- two-step algorithm-based approach (Experimental): Perform the laparoscopic biopsy as a discretion of attending physician's decision, but if the below conditions are met, do not perform the laparoscopic biopsy.
  1. Blood ELISPOT >= 6 spots or ascites adenosine deaminase > 20 IU/L, and
  2. Ascites ELISPOT/Blood ELISPOT rato > 3
  Interventions: Other: Blood and Ascites ELISPOT

INTERVENTIONS:
Other: Blood and Ascites ELISPOT
  Arms: two-step algorithm-based approach

SUMMARY:
The diagnosis of tuberculous peritonitis (TBP) is still challenging, and largely dependent on invasive procedures such as laparoscopy. A recently developed RD-1 gene-based assay for diagnosing TBP shows has given promising results. The investigators thus created a 2-step algorithm using the Blood/Ascites ELISPOT assays and adenosine deaminase (ADA) in ascites for differentiation of TBP from other diagnoses (Blood ELISPOT ≥6 spots or ADA ≥ 21 U/L' as a rule-out test and 'Ascites/Blood ratio ≥3' as a rule-in test). This study is the randomized controlled trial on whether this 2-step algorithm-based approach can reduce the laparoscopic biopsy for the diagnosis of TBP in patients with suspected TBP.

ELIGIBILITY:
Inclusion Criteria:

* all patients with suspected tuberculous peritonitis
* age 16 or more
* formal informed consent

Exclusion Criteria:

* not specified

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
the frequency of laparoscopic biopsy | 1 week after the enrollment

SECONDARY OUTCOMES:
the frequency of correct or wrong diagnosis | 6 months after the enrollment
  the frequency of correct or wrong diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Han Kim, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea